CLINICAL TRIAL: NCT00798772
Title: A Randomized Control Clinical Trial Of Micronutrient & Antioxidant Supplementation in Persons With Untreated HIV Infection
Brief Title: Micronutrients and Antioxidants in HIV Infection
Acronym: MAINTAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network); Ontario HIV Treatment Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTN 238
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: HIV Infection
Keywords: HIV infection; Micronutrients; Antioxidants
MeSH Terms: conditions — HIV Infections | interventions — Micronutrients; Antioxidants; Geritol; Minerals

STUDY DESIGN:
Intervention Model Description: Treatment group (Group A): Will receive micronutrients and antioxidants. Control group (Group B): Will receive identical appearing RDA multivitamins and minerals
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Broad spectrum micronutrients (Experimental): The experimental treatment medications (micronutrients and antioxidants) will be taken as one packet (8 capsules) twice a day with meals. Because of the presence of calcium, iron and zinc in the study medication, any other medication must be taken at least two hours before or after taking it. Participants may initiate the intervention at half dose (one packet of 8 capsules once a day) and increase to full dose after one week.
  The intervention will last for two years.
  Interventions: Dietary Supplement: Micronutrients and antioxidants
- B: Identical appearing multivitamins (Active Comparator): The active comparator/control medications (identical appearing RDA multivitamins and minerals) will be taken as one packet (8 capsules) twice a day with meals. Because of the presence of calcium, iron and zinc in the study medication, any other medication must be taken at least two hours before or after taking it. Participants may initiate the intervention at half dose (one packet of 8 capsules once a day) and increase to full dose after one week.
  The intervention will last for two years.
  Interventions: Dietary Supplement: Multivitamins and minerals

INTERVENTIONS:
Dietary Supplement: Micronutrients and antioxidants — 8 capsules twice daily for two years
  Other Names: K-PAX Ultra
  Arms: A: Broad spectrum micronutrients
Dietary Supplement: Multivitamins and minerals — 8 capsules twice daily for two years
  Other Names: Centrum-like multivitamins and minerals
  Arms: B: Identical appearing multivitamins

SUMMARY:
Infection with human immunodeficiency virus (HIV) causes decline in immunity or the ability to fight infection and progresses to acquired immunodeficiency disease (AIDS). Anti-HIV drug treatment has improved the prognosis of persons with HIV infection, but is expensive and potentially toxic. Low micronutrient levels occur in the blood even in early stages of HIV infection and increase risk of a poorer prognosis, but the role of micronutrient and antioxidant supplements in medical management of HIV/AIDS is not well defined. The proposed clinical trial aims to assess if supplementation of untreated HIV-infected adults with a micronutrient and antioxidant preparation can delay decline in immunity or disease progression or start of anti-HIV drug treatment compared with supplementation with standard multivitamins. If the findings are positive, the study has implications for health and health care savings.

DETAILED DESCRIPTION:
Background: Antiretroviral therapy (ART) has improved the prognosis of persons with human immunodeficiency virus (HIV) infection, but is expensive and potentially toxic. Micronutrient deficiencies occur even in early stages of HIV infection and increase risk of morbidity, disease progression to acquired immunodeficiency syndrome (AIDS) and mortality, but the role of micronutrient antioxidant supplements in medical management of HIV/AIDS is not clear.

Objective: To determine if supplementation of untreated asymptomatic HIV-infected persons with a broad-spectrum micronutrient and antioxidant preparation will reduce the rate of decline of CD4 T lymphocyte count, or delay emergence of documented CDC-defined AIDS-defining illness, or start of ART compared to 100% recommended daily allowance (RDA) multivitamins and minerals, and is safe.

Study design: A prospective, randomized, controlled, double blind clinical trial of supplementation of 218 untreated asymptomatic HIV-infected adults with a micronutrient and antioxidant preparation or identical appearing RDA multivitamins and minerals for two years, with quarterly follow up in clinic for assessment of time from baseline to CD4 count <350 mm3, or emergence of documented CDC-defined AIDS-defining illness, or start of ART.

Participants and sample size: 218 participants from clinics in Ontario and other participating centres of the CIHR Canadian HIV Trials Network (CTN).

Study duration: approximately five years, allowing for approximately three years for participant accrual and two years follow-up.

Eligibility criteria: The main eligibility criteria are:

• Asymptomatic HIV-infected adults at least 18 years of age

• CD4+ cells ≥375 and ≤750 cells/mm3

• No previous ART (excluding less than seven days and perinatal transmission prophylaxis) Study intervention: Oral supplementation with a broad spectrum micronutrient and antioxidant preparation (n=109) or identical appearing RDA multivitamins and minerals (n=109).

Primary outcome: Time from baseline to CD4+ cell count <350 cells/mm3 (confirmed by two measures at least one week apart), or emergence of documented CDC-defined AIDS-defining illness, or start of ART

Secondary outcomes:

• Non-AIDS related adverse events

• Tolerance of and adherence to study medication

• Time from baseline to CD4+ cell count <350 cells/mm3 (confirmed by two measures at least one week apart)

• Time from baseline to emergence of documented CDC-defined AIDS-defining illness

• Time from baseline to start of ART

• Serial quarterly lymphocyte measures: absolute lymphocyte count (ALC), CD4+, CD8+, and CD3+ cell counts, CD4%, CD8%, CD4:CD8

• Serial quarterly HIV RNA plasma viral load

• Serum chemistries: Glucose, BUN, creatinine, total protein, C-reactive protein, albumin, alkaline phosphatase, ALT, AST, total bilirubin

• Serum micronutrient levels: Carotene (quarterly) and vitamin B12 (quarterly), folate (six monthly) and vitamin D (25-OHD, six monthly)

• Quality of Life measures: MOS HIV, EuroQol, and Health Utilities Index (HUI) Statistical analysis: Analysis of the primary outcome by intention-to-treat will compare time from baseline to primary outcome. Interim analyses are planned once 100 participants are followed for one year.

ELIGIBILITY:
Inclusion Criteria:

* be an asymptomatic HIV infected adult
* at least 18 years of age
* have CD4+ cells between 375 and 750 cells/mm3
* have received no ART (excluding less than seven days and perinatal transmission prophylaxis)
* if a woman of child bearing potential, have a negative pregnancy test within two weeks prior to randomization and agree to practice barrier method of birth control during the study
* be willing and able to sign informed consent and to comply with the study protocol

Exclusion Criteria:

* have HIV-2 infection alone
* have known allergy or intolerance to any study medication ingredient
* be pregnant
* have active treatment for an acute opportunistic infection or malignancy
* have ALT greater than 3 x normal range
* have known cirrhosis of the liver
* have serum creatinine less than 133 umol/L
* abuse alcohol and recreational drugs
* be taking micronutrient (except vitamin D*) or natural health product supplements within 30 days of randomization *Maximum 2000 IU daily (Health Canada Guidelines).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2009-01; Primary Completion 2014-05 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Time from baseline to CD4+ cell count <350 cells/mm3 (confirmed by two measures at least one week apart), or emergence of documented CDC-defined AIDS-defining illness, or start of ART | Quarterly

SECONDARY OUTCOMES:
Non-AIDS related adverse events | Quarterly
Tolerance of and adherence to study medication | Quarterly
Time from baseline to CD4+ cell count <350 cells/mm3 (confirmed by two measures at least one week apart) | Quarterly
Time from baseline to emergence of documented CDC-defined AIDS-defining illness | Quarterly
Time from baseline to start of ART | Quarterly
Serial quarterly lymphocyte measures (ALC, CD4+, CD8+, and CD3+ cell counts, CD4%, CD8%, CD4:CD8) | Quarterly
Serial quarterly HIV RNA plasma viral load | Quarterly
Serum chemistries: Glucose, BUN, creatinine, total protein, albumin, alkaline phosphatase, ALT, AST, total bilirubin, | Quarterly
Serum micronutrient levels: carotene (quarterly), vitamin B12 (quarterly), folate (six monthly) and vitamin D (25-OHD six monthly) | Quarterly or as specified
Quality of Life measures | Quarterly

CONTACTS AND LOCATIONS:
Overall Officials: William Cameron, MD, FRCPC, Principal Investigator — University of Ottawa at The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Austin J, Singhal N, Voigt R, Smaill F, Gill MJ, Walmsley S, Salit I, Gilmour J, Schlech WF 3rd, Choudhri S, Rachlis A, Cohen J, Trottier S, Toma E, Phillips P, Ford PM, Woods R, Singer J, Zarowny DP, Cameron DW; CTN 091/CRIT Cartenoids Study Group. A community randomized controlled clinical trial of mixed carotenoids and micronutrient supplementation of patients with acquired immunodeficiency syndrome. Eur J Clin Nutr. 2006 Nov;60(11):1266-76. doi: 10.1038/sj.ejcn.1602447. Epub 2006 May 24. PMID 16721396
- [Background] Kaiser JD, Campa AM, Ondercin JP, Leoung GS, Pless RF, Baum MK. Micronutrient supplementation increases CD4 count in HIV-infected individuals on highly active antiretroviral therapy: a prospective, double-blinded, placebo-controlled trial. J Acquir Immune Defic Syndr. 2006 Aug 15;42(5):523-8. doi: 10.1097/01.qai.0000230529.25083.42. PMID 16868496
- [Derived] Wobeser WL, McBane JE, Balfour L, Conway B, Gill MJ, Huff H, Kilby DLP, Fergusson DA, Mallick R, Mills EJ, Muldoon KA, Rachlis A, Ralph ED, Rosenes R, Singer J, Singhal N, Tan D, Tremblay N, Vo D, Walmsley SL, Cameron DW; MAINTAIN Study Group. A randomized control trial of high-dose micronutrient-antioxidant supplementation in healthy persons with untreated HIV infection. PLoS One. 2022 Jul 14;17(7):e0270590. doi: 10.1371/journal.pone.0270590. eCollection 2022. PMID 35834528
- [Derived] Balfour L, Spaans JN, Fergusson D, Huff H, Mills EJ, la Porte CJ, Walmsley S, Singhal N, Rosenes R, Tremblay N, Gill MJ, Loemba H, Conway B, Rachlis A, Ralph E, Loutfy M, Mallick R, Moorhouse R, William Cameron D. Micronutrient deficiency and treatment adherence in a randomized controlled trial of micronutrient supplementation in ART-naive persons with HIV. PLoS One. 2014 Jan 21;9(1):e85607. doi: 10.1371/journal.pone.0085607. eCollection 2014. PMID 24465617